CLINICAL TRIAL: NCT06545747
Title: A Randomized Controlled Phase III Study of Adaptive Hypofractionated Radiotherapy Combined With Concurrent Chemotherapy and Consolidative Immunotherapy in Locally Advanced Non-Small Cell Lung Cancer Based on Dynamic Enhanced Magnetic Resonance Imaging
Brief Title: Adaptive Hypofractionated Radiotherapy for Locally Advanced NSCLC Based on Dynamic Enhanced MRI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2024-001
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: hypo-fractionated radiotherapy; consolidative immunotherapy; MRI-guided
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI-based hypo-RT (Experimental): Patients will receive split-course hypo-RT combined with concurrent chemotherapy and consolidative immunotherapy. The experimental arm will undergo adaptive dose-painting hypo-RT based on DCE-MRI.
  Interventions: Radiation: DCE-MRI based split-course hypo-RT; Drug: Concurrent chemotherapy; Drug: Consolidative immunotherapy
- CT-based hypo-RT (Active Comparator): Patients will receive split-course hypo-RT combined with concurrent chemotherapy and consolidative immunotherapy. The control arm will undergo hypo-RT based on CT.
  Interventions: Radiation: CT based split-course hypo-RT; Drug: Concurrent chemotherapy; Drug: Consolidative immunotherapy

INTERVENTIONS:
Radiation: DCE-MRI based split-course hypo-RT — Tumor delineation will be based on DCE-MRI and CT. MRI help define the tumor boundary. Different radiation doses will be delivered based on the Ktrans value of the tumor area on DCE-MRI.
  Arms: MRI-based hypo-RT
Radiation: CT based split-course hypo-RT — Tumor delineation will be based on CT. The total dose for both the first and boost courses of hypo-RT to the tumor area will be constant.
  Arms: CT-based hypo-RT
Drug: Concurrent chemotherapy — Concurrent Chemotherapy consists of weekly albumin-bound paclitaxel 50mg/m2, d1 plus cisplatin 25mg/m2，d1.
Drug: Consolidative immunotherapy — Consolidative PD-1/PD-L1 inhibitors

SUMMARY:
This study is a randomized phase III trial that aiming to investigate the role of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) guided hypofractionated radiotherapy (hypo-RT) in patients with locally advanced non-small cell lung cancer (LA-NSCLC) who are planned to receive hypo-RT combined with concurrent chemotherapy and consolidative immunotherapy. Patients will be randomized in a 1:1 ratio into two groups:

1. The study group will undergo adaptive dose-painting hypo-RT based on DCE-MRI.
2. The control group will undergo hypo-RT based on enhanced CT.

The treatment-related toxicity, local control and long-term survival will be evaluated compared between MRI-guided and CT-guided hypo-RT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 75 years old.
* Patients must have histological or cytological confirmation of locally advanced, unresectable (stage III) non-small cell lung cancer (NSCLC).
* No prior radiation therapy or surgery.
* Expected life expectancy of at least 12 weeks.
* World Health Organization (WHO) performance status score of 0 or 1.
* Able to undergo magnetic resonance imaging (MRI) examination.
* Organ and bone marrow function meeting the following criteria: Forced expiratory volume in 1 second (FEV1) ≥ 800 ml; Absolute neutrophil count ≥ 1.5 × 10^9/L; Platelets ≥ 100 × 10^9/L; Hemoglobin ≥ 9.0 g/dL; Serum creatinine clearance rate calculated by the Cockcroft-Gault formula ≥ 50 mL/min (Cockcroft and Gault 1976); Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN); Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN.

Exclusion Criteria:

* Contraindications to MRI examination.
* Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study.
* Histological type of mixed small cell and non-small cell lung cancer.
* Major surgery performed within 4 weeks prior to entering the study (excluding vascular access).
* History or occurrence of autoimmune disease within the past 2 years.
* Active or history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplantation requiring immunosuppressive therapy.
* Average QT interval (QTc) ≥ 470 ms calculated from 3 ECG cycles using Bazett's correction.
* Uncontrolled comorbidities, including but not limited to persistent or active infection, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmia, active peptic ulcer disease or gastritis, active bleeding disorder, human immunodeficiency virus (HIV), or psychiatric/social situations that would limit compliance with study requirements or impair the ability to provide written informed consent.
* Active tuberculosis.
* Receipt of a live attenuated vaccine within 30 days prior to the start of the study.
* History of another primary malignancy within 5 years, excluding adequately treated basal or squamous cell skin cancer or in situ cervical cancer.
* Pregnant or breastfeeding women; or males and females of reproductive potential not using effective contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
treatment-related G2+ respiratory toxicity | Recorded from the enrollment to 1 year after the completion of hypo-RT or 3 months after the completion of consolidative immunotherapy
  the percentage of patients who developed G2+ respiratory toxicity, including pneumonitis and proximal bronchial tree toxicity
progression-free survival rate | 2-year

SECONDARY OUTCOMES:
local control rate | 2-year
overall survival rate | 2-year
patient reported outcome assessed by QLQ-C30 | 2 year
  assessed by QLQ-C30
patient reported outcome | 2 year
  assessed by QLQ-LC13 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No